CLINICAL TRIAL: NCT06099990
Title: A Multicenter, Randomized, Double-blind Phase Ib/III Clinical Study of Dalpiciclib Isethionate Tablets Combined With Abiraterone Acetate Tablets (I) and Prednisone Tablets (AA-P) Versus Placebo Combined With AA-P in Treatment of High-volume, Metastatic, Hormone-sensitive Prostate Cancer (mHSPC).
Brief Title: Dalpiciclib Isethionate Tablets Combined With Abiraterone Acetate Tablets (I) and Prednisone Tablets (AA-P) Versus Placebo Combined With AA-P in Treatment of High-volume, Metastatic, Hormone-sensitive Prostate Cancer (mHSPC)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR6390-305
Record Dates: First submitted 2023-10-13; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: High-volume, Metastatic, Hormone-sensitive Prostate Cancer (mHSPC)
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dalpiciclib+ abiraterone+ prednisone (Experimental)
  Interventions: Drug: dalpiciclib isethionate tablets; abiraterone acetate tablets; prednisone tablets
- placebo+abirarerone+prenisone (Placebo Comparator)
  Interventions: Drug: placebo; abiraterone acetate tablets; prednisone tablets

INTERVENTIONS:
Drug: dalpiciclib isethionate tablets; abiraterone acetate tablets; prednisone tablets — dalpiciclib+ abiraterone+ prednisone
  Arms: dalpiciclib+ abiraterone+ prednisone
Drug: placebo; abiraterone acetate tablets; prednisone tablets — placebo+abirarerone+prenisone
  Arms: placebo+abirarerone+prenisone

SUMMARY:
This study was to evaluate the safety and efficacy of dalcilide tablets in combination with AA-P in the treatment of subjects with high tumor burden mHSPC and to determine the second stage starting dose and progression-free survival（rPFS） based on BICR assessment

ELIGIBILITY:
Inclusion Criteria:

1. Age of ≥ 18 years old,male
2. ECOG PS score of 0 or 1；
3. Prostate adenocarcinoma confirmed by histological。
4. ADT no more than 3 months prior to randomization (when docetaxel is not used) with no radiographic or PSA progression
5. Receiving or maintaining androgen deprivation therapy (ADT) during the planned study period, i.e. continuous treatment with luteinizing hormone-releasing hormone analogues (LHRHA) (drug castration) or prior bilateral orchiectomy (surgical castration)
6. Voluntarily participate in this clinical trial, understand the study procedure and have signed informed consent

Exclusion Criteria:

1. Previous ADT, chemotherapy, surgery, external radiation exposure, brachytherapy, radiopharmaceuticals, or experimental topical treatments (eg, radiofrequency ablation, cryoponic, high-energy focused ultrasound) for prostate cancer
2. Previous use of CDK4/6 inhibitors (such as piperaciclib, rebocillib and abeceptil), second-generation androgen receptor antagonists (such as enzalutamide, apatamide, darotamide, revilumide and proclomide, etc.), ketoconazole, abiraterone acetate or other investigational drugs that inhibit androgen synthesis (such as TAK-700), other anti-tumor biological therapy, targeted therapy or tumor immunotherapy
3. Confirmed by imaging, there are brain tumor foci
4. History of severe lung disease such as interstitial pneumonia
5. Plan to receive any other antitumor therapy during this trial
6. Inability to swallow, chronic diarrhea and intestinal obstruction, or other factors that affect drug taking and absorption

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Adverse event (AE) incidence | approximately 63 months

SECONDARY OUTCOMES:
PK： Steady-state trough concentrations of Dalsili and Abiraterone (Cmin, ss) | approximately 6 months
rPFS | approximately 63 months
  Time from randomisation to radiologically confirmed progressive disease or death due to any cause
PSA response rate | approximately 63 months
  In patients who had not started androgen deprivation prior to randomization, the proportion of patients whose PSA levels were ≥ 90% lower than baseline by the end of the study treatment week
ORR | approximately 63 months
  Objective response rate+ The proportion of participants evaluated according to RECIST v1.1 and PCWG3 criteria that achieved predetermined tumor volume reduction and maintained the minimum duration was the sum of the proportion of complete and partial responses
Time to PSA progression | approximately 63 months
  Time from randomisation to the first time of PSA progression

IPD SHARING:
Plan to Share IPD: Undecided